CLINICAL TRIAL: NCT05967286
Title: Olaparib Plus Low-Dose Alpelisib for Breast Cancer: A ComboMATCH Treatment Trial
Brief Title: Olaparib and Alpelisib for Treatment of Metastatic Breast Cancer, A ComboMATCH Treatment Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - Protocol moved to Withdrawn
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-05623; NCI-2023-05623 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-A2 (Other: Alliance for Clinical Trials in Oncology); EAY191-A2 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2023-07-28; First posted 2023-08-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic HER2-Negative Breast Carcinoma; Unresectable HER2-Negative Breast Carcinoma
MeSH Terms: interventions — Alpelisib; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Arm A (olaparib, alpelisib) (Experimental): Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Drug: Alpelisib; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Magnetic Resonance Imaging; Drug: Olaparib
- Cohort 2, Arm B (olaparib, alpelisib) (Experimental): Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Drug: Alpelisib; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: Positron Emission Tomography
- Cohort 2, Arm C (olaparib) (Active Comparator): Patients receive olaparib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients experiencing disease progression have the option to migrate to Cohort 3, Arm D. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib
- Cohort 3, Arm D (olaparib, alpelisib) (Experimental): Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Drug: Alpelisib; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Alpelisib — Given PO
  Other Names: BYL719; Phosphoinositide 3-kinase Inhibitor BYL719; Piqray; VIJOICE
  Arms: Cohort 1, Arm A (olaparib, alpelisib); Cohort 2, Arm B (olaparib, alpelisib); Cohort 3, Arm D (olaparib, alpelisib)
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scans
  Other Names: Bone Scintigraphy
  Arms: Cohort 1, Arm A (olaparib, alpelisib); Cohort 2, Arm C (olaparib); Cohort 3, Arm D (olaparib, alpelisib)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
  Arms: Cohort 2, Arm B (olaparib, alpelisib); Cohort 2, Arm C (olaparib); Cohort 3, Arm D (olaparib, alpelisib)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
  Arms: Cohort 2, Arm B (olaparib, alpelisib); Cohort 3, Arm D (olaparib, alpelisib)

SUMMARY:
This phase II ComboMATCH treatment trial studies the effect of adding a drug called BYL719 (alpelisib) to the usual treatment of olaparib in patients with breast cancer that has spread from where it first started (breast) to other places in the body (metastatic). Olaparib is an inhibitor of PARP, an enzyme that helps repair DNA when it becomes damaged. Blocking PARP may help keep tumor cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Alpelisib blocks certain proteins, which may help keep tumor cells from growing and may kill them. It is a type of kinase inhibitor. Giving alpelisib in combination with olaparib may be able to improve treatment results for patients with metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether BYL719 (alpelisib) and olaparib combination therapy improves progression-free survival (PFS) compared to olaparib alone in patients with PARP-inhibitor naive metastatic HER2-negative breast cancer. (Cohort 2) II. To determine the ORR of BYL719 (alpelisib) and olaparib in patients with PARP-inhibitor-resistant HER2-negative metastatic breast cancer. (Cohort 3)

SECONDARY OBJECTIVES:

I. To determine whether BYL719 (alpelisib) and olaparib combination therapy improves objective response rate (ORR), overall survival (OS), clinical benefit rate (CBR), and tolerability compared to olaparib alone in patients with PARP-inhibitor naive metastatic HER2-negative breast cancer. (Cohort 2) II. Collect tissue and provide it to the ComboMATCH Registration Protocol to assess concordance between the diagnostic tumor mutation profile generated by the Designated Laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) mutation profile from plasma, as described in ComboMATCH Registration Protocol. (Cohort 2) III. To assess the clinical activity of BYL719 (alpelisib) and olaparib combination therapy as measured by progression free survival (PFS), overall survival (OS), clinical benefit rate (CBR), and tolerability in patients with PARP-inhibitor-resistant HER2 negative metastatic breast cancer. (Cohort 3) IV. Collect tissue and provide it to the ComboMATCH Registration Protocol to assess concordance between the diagnostic tumor mutation profile generated by the Designated Laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment ctDNA mutation profile from plasma, as described in ComboMATCH Registration Protocol. (Cohort 3)

TRANSLATIONAL OBJECTIVES:

I. To explore the effect of PIK3CA mutations on ORR and PFS in the study population.

II. To assess correlates of response to olaparib and BYL719 (alpelisib) therapy in the study population including:

IIa. Germline and somatic mutations in DNA repair genes in blood and tumor samples from patients; IIb. DNA and ribonucleic acid (RNA) signatures, loss of heterozygosity (LOH) and other measures of tumor genomic loss and instability from unbiased sequencing of DNA and RNA from patients; IIc. Biomarkers of DNA repair defects or homologous recombination repair deficiency in tumor tissue (e.g. RAD51 nuclear foci); IId. Clinical factors (e.g. prior chemotherapy; estrogen receptor status of tumor).

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT 1: PARP-inhibitor naive patients are assigned to Arm A.

ARM A: Patients receive olaparib orally (PO) twice daily (BID) and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML). Patients also undergo magnetic resonance imaging (MRI), computed tomography (CT), and/or positron emission tomography (PET) scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

COHORT 2: PARP-inhibitor naive patients are randomized to 1 of 2 arms.

ARM B: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

ARM C: Patients receive olaparib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients experiencing disease progression have the option to migrate to Cohort 3, Arm D. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

COHORT 3: PARP-inhibitor resistant patients are assigned to Arm D.

ARM D: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

After completion of study treatment, patients are followed every 6 months for up to 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-A2 based on the presence of an actionable mutation as defined in EAY191
* Metastatic or unresectable breast cancer that is HER2-negative (by American Society of Clinical Oncology-College of American Pathologists [ASCO-CAP] guidelines)
* Patients with estrogen receptor positive (ER+) or ER-negative disease are eligible
* Germline or deleterious somatic mutation in at least one of: BAP1, BARD1, BRCA1, BRCA2, BRIP1 (FANCJ), FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11,PALB2, RAD50, RAD51B, RAD51C, RAD51D
* COHORTS 1 AND 2 (PARP-INHIBITOR NAIVE): No prior PARP-inhibitor is allowed. Prior mTOR- or AKT-inhibitor is allowed
* COHORTS 1 AND 2 (PARP-INHIBITOR NAIVE): PIK3CA mutation status
* COHORT 3 (PRIOR PARP-INHIBITOR): Patient must have received and progressed on prior PARP inhibitor therapy in any setting; intervening lines of therapy are allowed
* At least one measurable lesion that can be accurately assessed at baseline by CT (MRI where CT is contraindicated) and is suitable for repeated assessment as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Prior PI3K inhibitor therapy is allowed
* Patients with estrogen receptor positive (ER+) disease are eligible after progression on at least 1 prior endocrine treatment in the metastatic setting
* No treatment within 4 weeks of registration which includes: investigational medicinal product (IMP), systemic anti-cancer treatment (cytotoxic chemotherapy, immunotherapy, targeted therapy except for PI3K inhibitors, biologics, tumor embolization, or monoclonal antibodies). If there is a period needed for the IMP or systemic treatment to be cleared from the body that may take longer than 4 weeks (i.e. period of 5 half lives), the longer time period should be utilized
* No major surgery done =< 14 days prior to registration, or patients must have recovered from any effects from any major surgery that occurred > 14 days prior to registration
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown and an agent that has known genotoxic, mutagenic and teratogenic effects

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status =< 2 (or Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total Bilirubin =< 1.5 x upper limit of normal (ULN)

  * Except in the event of Gilbert disease, in which case total bilirubin must be =< 2 x ULN
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional ULN
* Hemoglobin (Hgb) >= 10.0 g/dL with no blood transfusion in the past 28 days
* Fasting plasma glucose (FPG) =< 140 mg/dL (7.7 mmol/L)
* Glomerular filtration rate (GFR) >= 50 mL/min

  * Based on a 24-hour urine test for creatinine clearance or estimated using the Cockcroft-Gault equation
* Patients must be able to swallow oral formulations of the agents and must not have gastrointestinal disorders likely to interfere with absorption of the study medication
* Patients must not have symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression are excluded unless considered to have received definitive treatment for this and evidence of clinically stable
* Patients with known myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML should be excluded
* Patients who have had previous organ transplant, allogeneic bone marrow transplant or double umbilical cord blood transplantation should be excluded
* Patients must not be considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with type 1 diabetes mellitus are not eligible. Those with controlled type 2 diabetes mellitus (T2DM) are eligible. Patients with controlled T2DM, including those on insulin treatment, must meet the fasting plasma glucose requirement
* Patients must not have a known hypersensitivity to olaparib or BYL719 (alpelisib)
* Patients must not have known active hepatitis (i.e., hepatitis B or C) or human immunodeficiency virus (HIV) with detectable viral load. Patients with a history of HIV with undetectable viral load within 6 months are eligible) as long as drug-drug interactions are safe with study drugs if on anti-retroviral treatment. Testing at baseline for hepatitis or HIV is recommended but not required. If a patient had a history of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated prior to registration. If a patient had a history of hepatitis C virus (HCV) infection, they must have received the appropriate treatment and have an undetectable HCV viral load prior to registration
* Patients must not have a Grade 2 neuropathy or greater, within 14 days prior to registration
* Chronic concomitant treatment with strong inhibitors of CYP3A4 (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) is not allowed on this study. Patients on strong or moderate CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study
* Chronic concomitant treatment with strong CYP3A4 inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil) is not allowed. Patients must discontinue 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents prior to registering to the study treatment
* Cohort Migration EAY191-A2 Eligibility Criteria: Patients treated with Cohort 2 control treatment olaparib who experience disease progression may elect to migrate to Cohort 3 and receive combination treatment with BYL719 (alpelisib) and olaparib. Patients who choose to do so must meet laboratory values and performance status requirements as above and must be begin treatment within 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-23 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (Cohort 2) | From randomization date until the time of disease progression or death due to any cause, assessed up to 5 years
  Will compare the PFS distributions between those treated with BYL719 (alpelisib) and olaparib versus (vs) olaparib. Despite this being a randomized phase II trial, we will utilize an intent to treat approach such that patients will be analyzed based on the treatment arm to which they were randomized. Will be compared between the two treatment arms using Kaplan-Meier methods. The hazard ratio, median PFS, and estimated PFS rates at 6, 12, 18, 24, and 30 months will be estimated along with corresponding 95% confidence intervals.
Objective response rate (ORR) (Cohort 3) | Up to 5 years
  Defined as the proportion of patients who documented a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 divided by the total number of evaluable patients in a cohort.

SECONDARY OUTCOMES:
ORR (Cohort 2) | Up to 5 years
  RECIST v1.1 criteria will be used to estimate ORR where ORR is defined as the number of evaluable patients achieving a response (PR or CR per RECIST v1.1) during treatment with study therapy divided by the total number of evaluable patients. Rates of response will be compared between treatment arms using a chi-square test (or Fisher's exact test as needed). Point estimates will be generated for objective response rates within each arm along with 95% confidence intervals using the Clopper-Pearson method.
PFS (Cohort 3) | From study entry to the first of either disease progression or death from any cause, assessed up to 5 years
  Disease progression will be determined based on RECIST 1.1 criteria. PFS will be estimated using the Kaplan-Meier method. The median PFS and corresponding 95% confidence interval will be reported. Patients will be censored at the last disease assessment date if they were alive and progression-free at the time of their last assessment. If a patient begins a non-protocol therapy, the patient will be censored at the last assessment date prior to start of non-protocol therapy.
Overall survival (OS) (Cohorts 2 and 3) | From registration until death due to any cause, assessed up to 5 years
  Patients who are alive at last follow-up will be censored at that time point. The distribution of OS will be estimated using method of Kaplan-Meier. The median OS and 95% confidence interval will be reported.
Clinical benefit rate (CBR) (Cohorts 2 and 3) | From registration until death due to any cause, assessed up to 5 years
  Defined as achieving CR, PR or stable disease (SD) while on treatment. Disease status will be assessed using RECIST v1.1 criteria. CBR will be calculated as the proportion of evaluable patients who achieve clinical benefit. The final CBR point estimate and corresponding 95% confidence interval will be calculated using Clopper-Pearson method.
Incidence of adverse events (Cohorts 2 and 3) | Up to 5 years
  All eligible patients that have initiated treatment will be considered evaluable for assessing AE rate(s). Patients will be evaluated for adverse events using the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AE(s) to the study treatment will be taken into consideration.
Concordance of diagnostic tumor mutation profile (Cohorts 2 and 3) | Up to 5 years
  Concordance of diagnostic tumor mutation profile generated by the Designated Laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment ctDNA mutation profile will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Gerburg M Wulf, Principal Investigator — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm